CLINICAL TRIAL: NCT05452694
Title: Pharmacogenetics and Pharmacokinetics of Oxycodone to Personalize Postoperative Pain Management Following Lumbar Spinal Fusion and Decompression Surgery in Adults
Brief Title: OpalGenix- Personalized Postoperative Pain Management Following Lumbar Spinal Fusion and Decompression Surgery in Adults
Status: Recruiting | Type: Observational
Sponsor: OpalGenix, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: STUDY22010019
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Lumbar Spine Stenosis; Lumbar Spine Degeneration
Keywords: Pain Management; Lumbar Spine Stenosis; Degenerative Lumbar Spine; Opioid Use
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — One blood collection will take place at the baseline visit consisting of 1 EDTA tube which will collect approximately 2-3mL. This blood collection will be used for genotyping CYP2D6.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The proposed research is an important extension of an ongoing perioperative personalized analgesia and intravenous opioid pharmacogenetic research. This research focuses on two of the most commonly used oral opioid analgesics, oxycodone, and methadone, in adults following lumbar spinal fusion and decompression surgery. Genetic signature and combinatorial pharmacogenetic approaches perform better than single-gene associations. This innovative translational research will for the first time evaluate simultaneously the effects of multiple genes and interactions on oxycodone and methadone's pharmacokinetics and optimal clinical dosing and on its safety and efficacy in the highly vulnerable pediatric population. This research's multigenetic signature findings can be easily extrapolated to adults undergoing surgery or using oxycodone and/or methadone for chronic and cancer pain and in identifying opioid abusers at risk of severe respiratory depression and death.

When methadone is given in addition to oxycodone for inpatient pectus excavatum repair and idiopathic scoliosis spinal fusions according to new departmental protocols, methadone pharmacokinetics and pharmacodynamics will also be evaluated.

DETAILED DESCRIPTION:
Multilevel lumbar spinal fusion and decompression surgeries (LSS) are common and extremely painful inpatient procedures associated with severe post-surgical pain, high incidence of CPSP, persistent and excessive opioid use, unsafe opioid prescribing and development of opioid use disorder (OUD), along with costly immediate postoperative opioid adverse events (AEs) and long hospital stays. Opioids are still widely used to manage acute surgical pain and remain a core component of multi-modal analgesic and enhanced recovery after surgery protocols (ERAS) for painful surgeries. About half of LSS patients suffer from uncontrolled severe surgical pain and significant adverse opioid effects due to opioids' narrow therapeutic indices and unpredictable inter-individual variations in pain perception and opioid responses. Risks associated with perioperative opioid use include immediate risks (life-threatening respiratory depression (RD), excessive sedation, postoperative nausea and vomiting (PONV), urinary retention, constipation, ileus and itching) that frequently delay recovery, require additional treatment or monitoring, increase cost of care, and prolong hospital stay. Long-term risks include opioid dependence, opioid-use disorder (OUD), and the consequent personal, financial and societal fall-out from opioid addiction.

While in the hospital, LSS patients report suboptimal surgical pain (and AEs) with short-acting opioids such as morphine, hydromorphone, and fentanyl. Post-discharge, despite receiving additional potent prescribed opioids such as oxycodone for >1-2 weeks at home, 20-50% of patients develop CPSP, largely due to suboptimal immediate surgical pain relief (the single greatest risk factor for CPSP). Patients who develop CPSP have high life-long risks for opioid use and misuse, contributing to the ongoing opioid epidemic and lost productive life. Poor surgical pain relief and opioid- AEs therefore result in negative consequences for patients, families, providers, and society, and constitute significant socio-economic burden. Thus, there is an urgent and unmet clinical need for a reliable and proactive tool to reduce opioid use and opioid-related AEs, enhance pain relief and prevent CPSP following painful surgeries.

CPSP is common following LSS: Effective and aggressive acute surgical pain management is critical to lower risks of developing CPSP. In a large prospective study assessing pain outcomes from 21 hospitals in 11 European countries (PAIN OUT cohort)120, 11.8% of patients reported moderate to severe CPSP at 12 months. The three risk factors for CPSP at 12 months, chronic preoperative pain, type of surgery and percentage of time in severe acute surgical pain, are very common in LSS patients. Importantly, orthopedic surgery is associated with 3-fold higher risk for CPSP compared with all other procedures. A 10% increase in the percentage of time in severe pain on the first postoperative day was associated with a 30% increase in the incidence of CPSP at 12 months (N=889). LSS is often associated with severe acute post-surgical pain, a high incidence of CPSP, excessive and persistent opioid use increasing cost of care significantly with high worker compensation costs with lost productivity. Thus, there is a clear need for more effective and safer pain management following LSS to prevent CPSP, risks of lost productivity, excessive opioid use, misuse, dependence and OUD.

High inter-individual variations in response to opioids can be explained by genetics and clinical risk factors, yet translational barriers prevent widespread adoption of genotype-guided care: Our many studies on genetic predictors of postoperative pain and opioid-related AEs, and published literature from other researchers demonstrate that genetic and clinical factors are associated with inter-individual variations in pain control and adverse outcomes with different opioids. Through genotype-based opioid selection, precision dosing and outpatient tailored opioid prescribing improve outcomes, there are many translational barriers. An important example is the use of CYP2D6 phenotyping to guide dosing or use of codeine, tramadol, hydrocodone, and oxycodone for improved safety and efficacy.

OpalGenix intends to revolutionize perioperative opioid and pain management with proactive and personalized risk prediction algorithms with >70% accuracy in predicting opioid AEs for precision pain and opioid management. GPS-Opioid will be a 510(k) cleared medical device that will enable preoperative genotyping of important and patented polygenetic markers shown to impact clinically and economically meaningful perioperative opioid and pain outcomes. The polygenetic markers predict opioid AEs better than single-gene associations: each gene, including CYP2D6, explains only 5-10% of clinical response variations while polygenetic models have >70% predictive accuracy as they combine important pharmacodynamics genes with well-known but less important genes involved in opioid metabolism such as CYP2D6. In addition, polygenetic models account for the synergistic effects of multiple risk alleles. Uniquely, GPS-Opioid also includes patented clinical risk factors with polygenetic signatures using a proprietary algorithm to identify patients at risk for experiencing uncontrolled severe pain, opioid-related AEs including RD and PONV, prolonged hospital stay, CPSP, opioid dependence and potential for developing OUD. Integration of GPS-Opioid in EHR, at the point-of-care, will enable perioperative clinicians with critical information they need to develop a personalized ERAS pain management plan prior to surgery to proactively minimize/eliminate costly opioid related adverse events, enhance surgical pain relief and avoid CPSP

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* American Society of Anesthesiologists (ASA) Physical Status 1, 2, or 3
* Undergoing lumbar spine surgeries (lumbar spine decompression, multilevel posterior spine fusion, internal fixation or a combination) for degenerative lumbar spine and lumbar spinal stenosis and requiring opioids for perioperative pain management

Exclusion Criteria:

* Children (<18 years of age)
* Pregnant women
* American Society of Anesthesiologists (ASA) Physical Status 4 or above
* Non-English speaking
* Outpatient surgery
* Concomitant additional surgical procedures
* Significant liver or kidney dysfunction
* Significant cardiorespiratory compromise
* Patients with polysubstance use (e.g., cocaine, marijuana, amphetamine, etc.)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will be adults undergoing lumbar spine surgeries that fit the inclusion criteria. Children will not be included as they are not seen at the specific site institution. Given the nature of the surgical procedure, pregnant women and women that may be pregnant will also not be included in this study population.
Sampling Method: Non-Probability Sample
Enrollment: 235 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-07-18 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Opioid-related Post-operative nausea and vomiting (PONV) | Post-operative up to 12 months
  PONV is measured with a binary yes/no response
Opioid-related sedation | Post-operative up to 12 months
  Sedation will be measured using the Riker Sedation Scale. The minimum score of 1 categorizes the patient as being unarousable, while the maximum score of 7 categorizes the patient as being dangerous agitation.
Opioid-related respiratory depression (RD) | Post-operative up to 12 months
  Respiratory depression is defined as abnormally slow respiratory rate which is below 12 breaths per minute. This will be measured with a binary yes/no response pulled from the electronic medical records.

SECONDARY OUTCOMES:
Opioid use | Pre-operative to post-operative up to 12-months
  Inpatient total opioid usage
Post-operative Pain Scores | Pre-operative to post-operative up to 12-months
  Pain scores will be measured using the patient-reported Numerical Rating Scale (NRS), in which a minimum score of 0 indicates no pain at all and a maximum score of 10 indicates the worst pain imaginable
Length of Hospital Stay | Post-operative day 1 up to 1-month
  Length of hospital stay will be recorded as the number of days a patient remained in the hospital post-operatively
Chronic Post-surgical Pain (CPSP) | Post-operative up to 12 months
  CPSP is defined as pain that develops after surgical invention and lasts at least 2 months. CPSP will be scored as yes/no.
Length of Prescribed Opioid Usage | Post-operative up to 12-months
  Length of prescribed opioid usage will be recorded as the number of days patient has an active prescription which will be obtained from electronic medical records
Opioid Dependence (OD) | Post-operative up to 12 months
  OD and OUD risk will be measured using the Current Opioid Misuse Measure (COMM) tool. The COMM is a 17-item questionnaire in which a score of 9 or higher is considered a positive screen for opioid misuse. Minimum score is 0 and maximum score is 68.
Opioid Use Disorder (OUD) Risk | Post-operative at 3-months
  OD and OUD risk will be measured using the Current Opioid Misuse Measure (COMM) tool. The COMM is a 17-item questionnaire in which a score of 9 or higher is considered a positive screen for opioid misuse. Minimum score is 0 and maximum score is 68.
Differences in fNIRS signals | Preoperative
  Differences in fNIRS task-based activations and resting state connectivity
QST Battery Responses | Preoperative
  Differences in responses to QST to characterize threshold and tolerance to cutaneous thermal and mechanical stimuli
Pain intensity scores after stair climbing task | Preoperative
  Verbal score from 0-100 on numeric rating scale (NRS) of pain following stair climbing task. Higher NRS scores indicate higher pain intensity.
Pain intensity scores after walking test | Preoperative
  Verbal score from 0-100 on NRS of pain following a 6-minute walking task. Higher NRS scores indicate higher pain intensity.
Duration of stair climbing task | Preoperative
  Differences in time taken to complete stair climbing task
Distance walked during 6-minute walking task | Preoperative
  Differences in distance walked during 6-minute walking task

CONTACTS AND LOCATIONS:
Overall Officials: Kathirvel Subramaniam, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (3):
- United States (3):
  - UPMC Montefiore Hospital, Pittsburgh, Pennsylvania
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC Pain Medicine at Centre Commons, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No